CLINICAL TRIAL: NCT03770286
Title: Treatment of Interproximal Carious Lesions on Primary Molar Teeth With SDF and Super Floss Application Versus SDF Without Super Floss Versus Fluoride Varnish Alone: a Pilot Phase 3 Randomized Controlled Trial
Brief Title: Treatment of Interproximal Cavities on Primary Molar Teeth With Silver Diamine Fluoride
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Los Angeles (Other)
Collaborators: University of Southern California (Other)
Responsible Party: Principal Investigator, alexander alcaraz, Medical Staff/USC Faculty CWR, Children's Hospital Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CHLA-18-00389
Record Dates: First submitted 2018-12-06; First posted 2018-12-10 (Actual); Results first posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-09

CONDITIONS: Dental Caries in Children; Dental Caries Class II; Dental Caries
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Intervention Model Description: Silver diamine fluoride is a medicament that can be used to remineralize and treat demineralized tooth structure. This studies Silver Diamine Fluoride application as a treatment for interproximal caries. It also compares Super Floss and Microbrush as ways in which to apply the medicament.
Who Masked: Outcomes Assessor
Masking Description: Evaluator of the x-rays will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Fluoride Varnish alone (Active Comparator): 5% sodium fluoride varnish will be applied to all teeth the day of acceptance into the study and then at 3 months, 6 months, and 12 months.
  Interventions: Device: 5% Fluoride Varnish
- SDF with Super Floss (Experimental): SDF will be applied to target interproximal lesions with the use of Super Floss for 1 minute. 5% sodium fluoride varnish will then be applied to all teeth. Both will occur the day of acceptance into the study and then at 3 months, 6 months, and 12 months.
  Interventions: Device: 5% Fluoride Varnish; Device: 38% Silver diamine fluoride; Device: Super Floss
- SDF without Super Floss (Experimental): SDF will be applied to around the (buccal, lingual, and occlusal) embrasures of the target interproximal lesions with the use of a microbrush for 1 minute. 5% sodium fluoride varnish will then be applied to all teeth. Both will occur the day of acceptance into the study and then at 3 months, 6 months, and 12 months.
  Interventions: Device: 5% Fluoride Varnish; Device: 38% Silver diamine fluoride

INTERVENTIONS:
Device: 5% Fluoride Varnish — Topical varnish
  Other Names: Voco ProFluorid Varnish
Device: 38% Silver diamine fluoride — Topical varnish
  Other Names: Advantage Arrest 38% Silver Diamine Fluoride; SDF
  Arms: SDF with Super Floss; SDF without Super Floss
Device: Super Floss — Floss will be used as a delivery agent of SDF to target interproximal carious lesion.
  Other Names: Oral-B Super Floss; woven floss; spongy floss
  Arms: SDF with Super Floss

SUMMARY:
This study investigates whether 1) Silver diamine fluoride (SDF) application using Super Floss can arrest and/or reverse initial interproximal caries on primary molars and 2) whether SDF applied with Super Floss is more effective in arresting or remineralizing initial interproximal lesion in comparison to SDF applied without Super Floss or fluoride varnish applied alone.

DETAILED DESCRIPTION:
Interproximal carious lesions are challenging to control and arrest due to difficulty reaching the contact area (in between teeth), limited salivary access, and poor flossing compliance in children and adolescents when flossing themselves. The vast majority of caries observed in children ages 5 to 10 are on interproximal surfaces.

Silver diamine fluoride (SDF) is a topical medicament touted as a very safe and noninvasive alternative and/or adjunct to topical fluoride treatment or restorative treatment to halt the progress ("arrest") of caries. SDF has been shown to remineralize ("reverse") demineralized enamel or dentin, inhibit collagenases to protect dentin collagen from destruction, and have bactericidal properties to cariogenic bacteria including streptococcus mutans. Normally, SDF is applied with a microbrush directly on an exposed carious lesion, but due to difficulty reaching interproximal carious lesions, an absorbent type of floss such as Super Floss has been proposed as a delivery method for SDF application.

The purpose of this study is to investigate whether 1) SDF application using Super Floss can arrest and/or reverse initial interproximal caries on primary molars and 2) whether SDF applied with Super Floss is more effective in arresting or remineralizing initial interproximal lesion in comparison to SDF applied without Super Floss or Fluoride varnish applied alone.

The study population includes healthy children, aged 3-12, with initial interproximal decay on deciduous molars identified by radiographs. In this study, initial decay is defined as radiographic decay within enamel or extending to the dentin-enamel junction based on International Caries Classification and Management System (ICCMS). Any eligible participant will be randomly allocated to one of three treatments: Fluoride varnish (Control) application alone versus SDF application without Super Floss (Control) versus SDF application with Super Floss (Intervention), which will be applied at the initial visit. At 3, 6, and 12 months, the participants will return for reapplication of their respective treatments. At the 6 month and 12 month mark, bitewing radiographs will be taken to determine status of the interested lesion(s). If a lesion progresses beyond the outer 1/3 of dentin, then the patient will be withdrawn and recommended routine restorative dental treatment. If a lesion arrests or reverses, then the current treatment will continue until end of study duration (12 months) and re-evaluated.

A statistician will be assisting us with descriptive statistics, cluster-adjusted chi-squared test, and other statistics to determine if any correlation exists.

ELIGIBILITY:
Inclusion Criteria:

* ASA I and ASA II children, aged 3-12
* Behavior of 3 or 4 on Frankl scale
* Radiographic decay within enamel or extending to the dentin-enamel junction based on International Caries Classification and Management System (ICCMS) Categories 1, 2 and 3 "Initial stages".
* Target interproximal lesion does not have existing restoration, recurrent decay, or adjacent teeth with existing restorations.

Exclusion Criteria:

* Children who are not ASA I or ASA II
* Children who are allergic to or intolerant of SDF
* Children who have known sensitivity to silver or heavy metal-ions, or have abnormal skin sensitization.
* Children who have ulcerative gingivitis or stomatitis.
* Carious interproximal lesions on primary molars in ICCMS Category 4, 5, or 6 18 , which signify the extent of the carious lesion radiographically reaching the middle 1/3 of dentin, inner 1/3 of dentin, and into the pulp respectively.
* Behavior of a child within the Frankl 1 or 2 category, indicating a "Definitely Negative" and "Negative" behavior, which may compromise safe application of SDF.

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 51 (Actual)
Dates: Start 2019-01-22 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Alcaraz, DDS, Principal Investigator — CHLA, USC
Locations (1):
- Childrens Hospital Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Horst JA, Ellenikiotis H, Milgrom PL. UCSF Protocol for Caries Arrest Using Silver Diamine Fluoride: Rationale, Indications and Consent. J Calif Dent Assoc. 2016 Jan;44(1):16-28. PMID 26897901
- [Background] Rosenblatt A, Stamford TC, Niederman R. Silver diamine fluoride: a caries "silver-fluoride bullet". J Dent Res. 2009 Feb;88(2):116-25. doi: 10.1177/0022034508329406. PMID 19278981
- [Background] Sihra R, Schroth RJ, Bertone M, Martin H, Patterson B, Mittermuller BA, Lee V, Patterson B, Moffatt ME, Klus B, Fontana M, Robertson L. The Effectiveness of Silver Diamine Fluoride and Fluoride Varnish in Arresting Caries in Young Children and Associated Oral Health-Related Quality of Life. J Can Dent Assoc. 2020 Jun;86:k9. PMID 32543369
- [Background] Hammersmith KJ, DePalo JR, Casamassimo PS, MacLean JK, Peng J. Silver Diamine Fluoride and Fluoride Varnish May Halt Interproximal Caries Progression in the Primary Dentition. J Clin Pediatr Dent. 2020;44(2):79-83. doi: 10.17796/1053-4625-44.2.2. PMID 32271666
- [Background] Schwendicke F, Meyer-Lueckel H, Stolpe M, Dorfer CE, Paris S. Costs and effectiveness of treatment alternatives for proximal caries lesions. PLoS One. 2014 Jan 27;9(1):e86992. doi: 10.1371/journal.pone.0086992. eCollection 2014. PMID 24475208

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were offered enrollment upon radiographic ID of qualifying lesions and meeting inclusion criteria.
Units Other Than Participants: Number of teeth with lesions
Period: Overall Study
Arm/Group | Fluoride Varnish Alone | SDF With Super Floss | SDF Without Super Floss
Started | 17; 60 Number of teeth with lesions (Units are described as teeth with lesions) | 17; 74 Number of teeth with lesions | 17; 81 Number of teeth with lesions
Completed | 10; 24 Number of teeth with lesions | 13; 33 Number of teeth with lesions | 12; 30 Number of teeth with lesions
Not Completed | 7; 36 Number of teeth with lesions | 4; 41 Number of teeth with lesions | 5; 51 Number of teeth with lesions
Not completed — Lost to Follow-up | 6 | 4 | 3
Not completed — Protocol Violation | 1 | 0 | 2

BASELINE CHARACTERISTICS:
Population: Ethnicity and gender were not collected
Units Other Than Participants: Teeth
Groups:
- Total: Total of all reporting groups
Arm/Group | Fluoride Varnish Alone | SDF With Super Floss | SDF Without Super Floss | Total
Number analyzed (Participants) | 10 | 13 | 12 | 35
Number analyzed (Teeth) | 24 | 33 | 30 | 87
Age, Categorical [Count of Participants; unit: Participants] — All participants are under the age of 18. Therefore, there are '0' in the categories of 18-65 and over 65.
  Participants
    <=18 years | 10 | 13 | 12 | 35
    Between 18 and 65 years | 0 | 0 | 0 | 0
    >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 6.5 (1.8) | 6.8 (1.7) | 6.2 (2.0) | 6.5 (1.8)
Sex: Female, Male [Count of Participants; unit: Participants] — Data was not collected on gender Population: Gender was not collected
  Participants
    number analyzed (Participants) | 0 | 0 | 0 | 0
    Female |  |  |  | 0
    Male |  |  |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Race/ ethnicity was not collected
  Participants
    number analyzed (Participants) | 0 | 0 | 0 | 0
    American Indian or Alaska Native |  |  |  | 0
    Asian |  |  |  | 0
    Native Hawaiian or Other Pacific Islander |  |  |  | 0
    Black or African American |  |  |  | 0
    White |  |  |  | 0
    More than one race |  |  |  | 0
    Unknown or Not Reported |  |  |  | 0

OUTCOME MEASURES:

1. Primary Outcome: Interproximal Caries Zone of Radiolucency
Description: Bitewing radiographs will be taken of target lesions at Day 1 (baseline). Target interproximal carious lesion(s) will be rated based on the zone of radiolucency on the radiographs using the International Caries Classification and Management System (ICCMS).
  Category 1 = Progression Category 2 = Stabilization Category 3 = Remineralization
Time Frame: Baseline to 6 months
Population: Total number of teeth
Measure: Number; unit: Number of teeth
Units Other Than Participants: Teeth
Arm/Group | Fluoride Varnish Alone | SDF With Super Floss | SDF Without Super Floss
Number analyzed (Participants) | 10 | 13 | 12
Number analyzed (Teeth) | 31 | 43 | 44
Number of teeth
  Category 1 = Progression | 9 | 7 | 10
  Category 2 = Stabilization | 12 | 31 | 22
  Category 3 = Remineralization | 10 | 6 | 11

2. Primary Outcome: Interproximal Caries Zone of Radiolucency
Description: Bitewing radiographs will be taken of target lesions at 6 months and compared. Target interproximal carious lesion(s) will be rated based on the zone of radiolucency on the radiographs using the International Caries Classification and Management System (ICCMS).
  Category 1 = Progression Category 2 = Stabilization Category 3 = Remineralization
Time Frame: 6 months to 12 months
Measure: Number; unit: Number of teeth
Units Other Than Participants: Teeth
Arm/Group | Fluoride Varnish Alone | SDF With Super Floss | SDF Without Super Floss
Number analyzed (Participants) | 10 | 13 | 12
Number analyzed (Teeth) | 12 | 19 | 21
Number of teeth
  Category 1 = Progression | 6 | 3 | 9
  Category 2 = Stabilization | 3 | 13 | 10
  Category 3 = Remineralization | 3 | 3 | 2

3. Primary Outcome: Interproximal Caries Zone of Radiolucency
Description: Bitewing radiographs will be taken of target lesions at 12 months and compared. Target interproximal carious lesion(s) will be rated based on the zone of radiolucency on the radiographs using the International Caries Classification and Management System (ICCMS).
  Category 1 = Progression Category 2 = Stabilization Category 3 = Remineralization
Time Frame: Baseline to 12 months
Measure: Number; unit: Number of teeth
Units Other Than Participants: Teeth
Arm/Group | Fluoride Varnish Alone | SDF With Super Floss | SDF Without Super Floss
Number analyzed (Participants) | 10 | 13 | 12
Number analyzed (Teeth) | 24 | 33 | 30
Number of teeth
  Category 1 = Progression | 8 | 8 | 10
  Category 2 = Stabilization | 10 | 20 | 13
  Category 3 = Remineralization | 6 | 5 | 7

ADVERSE EVENTS:
Time Frame: No SAEs or AEs were collected or monitored
Description: No SAEs or AEs were collected or monitored
Groups:
- Fluoride Varnish Alone; SDF With Superfloss; SDF Without Superfloss: No SAEs or AEs were collected or monitored.
Arm/Group | Fluoride Varnish Alone | SDF With Superfloss | SDF Without Superfloss
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
The study suffered from a small sample size and a considerable number of patients who missed follow-up visits. Higher than expected lack of treatment adherence can be attributed to the study being conducted amidst the challenging circumstances of the COVID-19 pandemic, which posed difficulties in ensuring consistent patient follow-ups and strict adherence to treatment timelines.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-07-31): https://cdn.clinicaltrials.gov/large-docs/86/NCT03770286/Prot_SAP_000.pdf